CLINICAL TRIAL: NCT00916734
Title: Assessing Patient Response to Therapeutic Exercise Based on the Clinical Prediction Rule for Spinal Manipulation
Brief Title: Assessing Patient Response to Therapeutic Exercise Based on Clinical Prediction Rule (CPR) for Spinal Manipulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daemen College (Other)
Responsible Party: Principal Investigator, Ronald J. Schenk, Associate Professor Physical Therapy, Daemen College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SOCH/IRB/0614
Record Dates: First submitted 2009-06-08; First posted 2009-06-09 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Low Back Pain
Keywords: McKenzie; thrust manipulation; clinical prediction rule
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Manipulation Group (Experimental): Subjects who received spinal thrust manipulation as an intervention.
  Interventions: Procedure: Spinal thrust manipulation
- McKenzie MDT Group (Active Comparator)
  Interventions: Procedure: MDT (McKenzie Method)

INTERVENTIONS:
Procedure: MDT (McKenzie Method) — Subjects who perform exercises in their direction of preference.
  Other Names: functional outcomes
  Arms: McKenzie MDT Group
Procedure: Spinal thrust manipulation — Subjects who receive spinal thrust manipulation as an intervention.
  Arms: Spinal Manipulation Group

SUMMARY:
The purpose of this study is to determine whether patients who meet the criteria of the clinical prediction rule for spinal manipulation may respond more favorably to repeated exercises according to a direction of preference (what makes the symptoms decrease). The investigators do not know which of these two commonly-used treatments (manipulation or specific exercise) is better to treat low back pain.

DETAILED DESCRIPTION:
With the trends in health care focusing on treatment effectiveness, it is important for physical therapists to select the most appropriate intervention according to patient classification. Physical therapy interventions for management of LBP include therapeutic exercises and spinal manipulation.

The purpose of this study is to determine whether patients who fit the Clinical Prediction Rule (CPR) for spinal manipulation may respond instead to exercise according to repeated lumbar movements in the direction of preference.

The subjects for this study will be comprised of individuals referred for treatment of low back pain and data will be collected by physical therapists with certification in MDT who had experience treating patients through the use of spinal manipulation. Patient functional questionnaires and impairment measures will be used to analyze the patient's perceived level of function and outcome.

Following the completion of an informed consent, subjects will undergo a physical therapy examination by a licensed physical therapist. Patients will be included in the study if they meet the CPR for spinal manipulation as describe in earlier research 6,11. Following the examination, all qualified subjects will be randomly assigned to either the (1) spinal manipulation group or (2) the McKenzie (MDT) group and will receive treatment in accordance with their assigned group. The assessment tools administered at the initial examination will be readministered for follow-up analysis.

ELIGIBILITY:
Inclusion Criteria:

* people who meet the clinical prediction rule for spinal manipulation

Exclusion Criteria:

* people receiving worker's compensation
* those who have had spinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain level as measured on numerical pain rating scale | 1 year

SECONDARY OUTCOMES:
Oswestry score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Schenk, PT, PhD, Principal Investigator — Daemen College
Locations (1):
- Daemen College, Amherst, New York, United States